CLINICAL TRIAL: NCT01794403
Title: A Randomized Study of Radiation Hypofractionation Via Extended Versus Accelerated Therapy (HEAT) For Prostate Cancer
Brief Title: Radiation Hypofractionation Via Extended Versus Accelerated Therapy (HEAT) For Prostate Cancer
Acronym: HEAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Jay L. Friedland MD Prostate Cancer Research Fund (Unknown)
Responsible Party: Principal Investigator, Matthew Abramowitz, MD, Assistant Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20110491; NCI-2019-06935 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP))
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: Radiation Therapy; Hypofractionation Radiotherapy; Extended Hypofractionation Radiotherapy; Accelerated Hypofractionation Radiotherapy; AHRT; EHRT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Extended Hypofractionation Radiotherapy (EHRT) Group (Experimental): Participants in this group will receive the EHRT intervention over a period of 6 weeks.
  Interventions: Radiation: Extended Hypofractionation Radiotherapy
- Accelerated Hypofractionation Radiotherapy (AHRT) Group (Experimental): Participants in this group will receive the AHRT intervention over a period of 2 weeks.
  Interventions: Radiation: Accelerated Hypofractionation Radiotherapy

INTERVENTIONS:
Radiation: Extended Hypofractionation Radiotherapy — A total dose of 70.2 Gy will be delivered in 26 fractions, 2.7 Gy to the Planning Target Volume (PTV) by Intensity Modulated Radiotherapy (IMRT) with stationary gantry or rotating gantry technique.
  Other Names: EHRT
  Arms: Extended Hypofractionation Radiotherapy (EHRT) Group
Radiation: Accelerated Hypofractionation Radiotherapy — A total dose of 36.25 Gy will be delivered in 5 fractions, 7.25 Gy each to the Planning Target Volume (PTV), by Stereotactic Body Radiotherapy (SBRT) techniques.
  Other Names: AHRT
  Arms: Accelerated Hypofractionation Radiotherapy (AHRT) Group

SUMMARY:
Accelerated Hypofractionation Radiotherapy for prostate cancer of 36.25 Gy delivered in 5 fractions will not be inferior to the standard treatment of 70.2 Gy given in 26 fractions with respect to four-year biochemical failure (PSA failure) by Phoenix definition post-treatment completion.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven prostate adenocarcinoma.

   * Gleason score 2-7 (reviewed by reference lab at UM).
   * Biopsy within one year of date of enrollment.
2. Clinical stage ≤ T2 based on DRE and/or ≤ T3a based on MRI (if done); N0-Nx; M0-Mx (AJCC 7th Edition)

   * T-stage and N-stage determined by physical exam and available imaging studies (CT, and/or MRI of the pelvis; see section 4.5). For MRI, questionable extracapsular extension is permitted. To distinguish blood from tumor the ideal study would be to acquire T2, T1 noncontrast and T1 dynamic contrast enhanced sequence, although this is not required. A small amount of extracapsular extension is permitted, as long as it can be included in the clinical target volume (CTV) and the constraints are met.
   * M-stage determined by physical exam, CT or MRI. Bone scan not required unless clinical findings suggest possible osseous metastases.
3. Prostate-Specific Antigen (PSA) < 20 ng/ml, obtained no greater than 3 months prior to enrollment.
4. Patients belonging in one of the following risk groups:

   * Low:

     * Clinical stage* T1-T2; Gleason ≤ 6, PSA ≤ 10 & <50% biopsy cores positive.
   * Intermediate:

     * Clinical stage T2b-T2c; Gleason ≤ 6, PSA ≤ 10 & <50% biopsy cores positive.
     * Clinical stage T1-T2; Gleason ≤ 6, PSA ≤ 10 & ≥50% biopsy cores positive.
     * Clinical stage T1-T2; Gleason = 7, PSA ≤ 10 & <50% biopsy cores positive or T1-T2; Gleason ≤ 6 & PSA >10 and < 20 & < 50% biopsy cores positive.
     * MRI stage T3a with evidence of extraprostatic extension is allowed.
     * Clinical stage is based on digital rectal exam (DRE). Seminal vesicle invasion on MRI is not eligible. T1a should be permitted if subsequent peripheral zone biopsies show tumor.
5. Prostate volume: ≤ 80 cc.

   * Determined using: volume = π/6 x length x height x width.
   * Measured from CT or MRI ≤90 days prior to enrollment.
6. Zubrod performance status 0-1.
7. No prior total prostatectomy or cryotherapy of the prostate.

   * Prior suprapubic prostatectomy, transurethral resection and laser ablation are permitted.
8. No prior radiotherapy to the prostate or lower pelvis.
9. No implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery, in the investigator's opinion.
10. No chemotherapy for a malignancy in the last 5 years.
11. No history of an invasive malignancy (other than this prostate cancer, or nonmetastatic basal or squamous skin cancers) in the last 5 years.
12. 4-6 months of androgen deprivation therapy (ADT) are allowed for intermediate risk patients. This must be declared prior to randomization. This may not have been started more than 2 months prior to randomization.
13. Patient must be able to have gold fiducial markers placed in the prostate (if on anticoagulants, must be cleared by a primary care physician or cardiologist), or if patient already has fiducial marker placed, they must be in accordance with the protocol specifications. Note: If a method of intrafraction prostate tracking is available which does not require fiducial markers, this will be adequate for this trial (i.e. fourth dimensional (4D) transperitoneal ultrasound, onboard MRI guidance).
14. Ability to understand and the willingness to sign a written informed consent document.
15. Willingness to fill out quality of life/psychosocial forms.
16. Age >= 35 and =< 85 years.
17. International Prostate Symptom Index (IPSS) (AUA) score ≤12

Exclusion Criteria:

1. Does not have a diagnosis of prostate adenocarcinoma.
2. Patient has clinical T3a or any evidence of T3b disease.
3. Patient has stage N1 or M1 disease.
4. Patients has a PSA of greater than 20 ng/ml, obtained no greater than 3 months prior to randomization.
5. Patient does not meet any of the risk groups outlined in section 3.1.4.
6. Prostate volume greater than 80 cc.
7. Zubrod performance status 2 or greater.
8. Prior total prostatectomy.
9. Prior radiation therapy to the prostate or lower pelvis.
10. Implanted hardware which limits treatment planning or delivery (determined by the investigator).
11. Chemotherapy within the past 5 years.
12. Diagnosis of an invasive malignancy within 5 years (other than current prostate cancer or non-metastatic basal or squamous skin cancers or non-metastatic curatively treated papillary thyroid carcinoma).
13. The use of more than 2 months of androgen deprivation therapy (ADT) prior to randomization, or plans for ADT to be continued for greater than 6 months.
14. Inability to have gold fiducial markers placed in the prostate, or fiducial markers already placed that are not in accordance with the protocol (Section 4.2.2). Note: If a method of intrafraction prostate tracking is available which does not require fiducial markers, this will be adequate for this trial (i.e. 4D transperitoneal ultrasound, onboard MRI guidance).
15. Unwilling or inability to give informed consent.
16. Not willing to fill out quality of life/psychosocial questionnaires.
17. IPSS score > to 12.
18. Age < 35 and > 85 years.

Ages: 35 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2013-04-04 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Achieving Four-Year Biochemical Failure. | Up to 4 years (After Completion of Intervention)
  The number of participants achieving four-year biochemical failure between both treatment arms will be reported. Biochemical Failure will be evaluated using the Phoenix definition wherein failure occurs when the Prostate Specific Antigen (PSA) is ≥ 2 ng/ml more than the lowest PSA measurement before the current one.

SECONDARY OUTCOMES:
Number of Participants Achieving Two-Year Failure. | Up to 2 years (After Completion of Intervention)
  The number of participants achieving either biochemical or clinical failure or positive biopsy. Biochemical Failure will be evaluated using the Phoenix definition wherein failure occurs when the Prostate Specific Antigen (PSA) is ≥ 2 ng/ml more than the lowest PSA measurement before the current one. Clinical failure will be reported as any clinical evidence of local progression or recurrence. A positive biopsy will be concluded via histological evaluation.
Number of Participants Experiencing Acute Treatment-Related Toxicity | Up to 5 months (After Completion of Intervention)
  Acute treatment-related toxicity will be reported as the number of participants experiencing treatment-related grade 3 or higher gastrointestinal (GI) or genitourinary (GU) adverse events during treatment or within three (3) months after treatment completion. Toxicity will be assessed using the descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Prostate Cancer Mortality Rate as Measured by Number of Deaths | Up to 5.25 years (After Completion of Intervention)
  The prostate cancer mortality rate will be reported as the number of deaths related to prostate cancer among participants.
Overall Survival | Up to 5.25 years (After Completion of Intervention)
  Overall survival will be reported as the elapsed time in months from randomization to death from any cause. For surviving patients, follow-up will be censored at the date of last contact.
Numbers of Participants Achieving ASTRO Consensus Definition (ACD) of Biochemical Failure | Up to 5.25 years (After Completion of Intervention)
  The number of participants achieving American Society for Therapeutic Radiation and Oncology (ASTRO) Consensus Definition (ACD) of biochemical failure will be reported. ACD failure is defined as three consecutive rises in post-treatment PSA, measured at the specified follow-up intervals.
HRQOL as Assessed by MAX-PC questionnaire | Up to 5.25 years (After Completion of Intervention)
  Health-related quality of life (HRQOL) will be measured using the scores on the Modified 18-item Memorial Anxiety Scale for Prostate Cancer (MAX-PC) from pre-treatment to post-treatment. The scale consists of 18 items (e.g. "I thought about prostate cancer even though I didn't mean to.") scored on a scale from 0 ("not at all") to 3 ("often"). Total scores range from 0 to 54, with higher scores indicating higher levels of anxiety.
HRQOL as Assessed by EPIC-Short Form-12 questionnaire | Up to 5.25 years (After Completion of Intervention)
  Health-related Quality of Life (HRQOL) will be measured using the Expanded Prostate Cancer Index Composite and Medical Outcomes Study Short Form-12 (EPIC-Short Form-12) to evaluate patient function and satisfaction after prostate cancer treatment. The questionnaire has 5 subscales (Urinary Function, Urinary Symptoms, Bowel Habits, Sexual Function and Hormonal Function). Each subscale has a total score ranging from 0-100, with higher scores representing better HRQOL.
Number of Participants Experiencing Late Treatment-Related Toxicity | Up to 5.25 years (After Completion of Intervention)
  Late treatment-related toxicity will be reported as the number of participants experiencing treatment-related grade 2 or higher gastrointestinal (GI) or genitourinary (GU) adverse events occurring more than three months after treatment completion. Toxicity will be assessed using the descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Percentage of Participants Achieving Efficacy | Up to 2 years (After Completion of Intervention)
  Efficacy will be reported as the percentage of participants achieving biochemical or clinical failure between participants with low and early intermediate risk for prostate cancer. Biochemical Failure will be evaluated using the Phoenix definition wherein failure occurs when the Prostate Specific Antigen (PSA) is ≥ 2 ng/ml more than the lowest PSA measurement before the current one. Clinical failure will be reported as any clinical evidence of local progression or recurrence.
Average Incremental Cost Utility Score as Measured by Quality Adjusted Life Years (QALYs) | Up to 5.25 years (After Completion of Intervention)
  An average cost utility score per patient for each treatment arm (AHRT and EHRT) will be reported as the quality adjusted life years among participants for that treatment. Cost utility will be calculated via analysis of the costs of a given treatment and compared to the cost utility of competing treatment.
Percentage of Participants with Residual Tumor Post-Treatment | 2.25 years
  The percentage of participants with residual tumor on both arms will be reported. The investigators will obtain prostate tissue from participants via biopsy two years after completion of protocol tissue. Tissue will analyzed for the expression of prostate cancer biomarkers. The expression of biomarkers in the post-treatment biopsies will be compared to that in the pre-treatment prostate biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Abramowitz, MD, Principal Investigator — University of Miami; Alan Pollack, MD, PhD, Principal Investigator — University of Miami
Locations (3):
- University of Miami, Miami, Florida, United States
- Northern Sydney Local Health District - Royal North Shore Hospital, St Leonards, New South Wales, Australia
- A.O.U. Città della Salute e della Scienza di Torino - University Hospital Trust of Turin, Turin, Turin, Italy

IPD SHARING:
Plan to Share IPD: No